CLINICAL TRIAL: NCT00613717
Title: Timing, Duration and Severity of Infant Iron Deficiency: Developmental Impacts
Brief Title: Healthy Infant Development Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01HD052069-01A2 (NIH); 1R01HD052069-01A2 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-03

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency
Keywords: iron deficiency anemia; iron deficiency; infant; development; behavior
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Behavior | interventions — Folic Acid; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- a (Experimental): pre- and early postnatal iron
  Interventions: Dietary Supplement: folic acid + iron prenatally, vits A & D + iron postnatally
- b (Experimental): iron prenatal only
  Interventions: Dietary Supplement: folic acid + iron prenatally, vitamins A & D postnatally
- c (Experimental): iron early postnatal only
  Interventions: Dietary Supplement: folic acid prenatally, vitamins A & D + iron postnatally
- d (Active Comparator): no iron pre- or postnatal
  Interventions: Dietary Supplement: folic acid prenatally, vitamins A & D postnatally

INTERVENTIONS:
Dietary Supplement: folic acid + iron prenatally, vits A & D + iron postnatally — Prenatally: pills by mouth, one per day, from the first prenatal visit until delivery, 400 mcg folic acid, 30 mg Fe.
  Postnatally: liquid by mouth, once per day, from 6 weeks old until 9 months old, 1 mg/kg/day Fe, 1500 IU vitamin A, 500 IU vitamin D.
  Arms: a
Dietary Supplement: folic acid + iron prenatally, vitamins A & D postnatally — Prenatally: pills by mouth, one per day, from the first prenatal visit until delivery, 400 mcg folic acid, 30 mg Fe.
  Postnatally: liquid by mouth, once per day, from 6 weeks old until 9 months old, 1500 IU vitamin A, 500 IU vitamin D.
  Arms: b
Dietary Supplement: folic acid prenatally, vitamins A & D + iron postnatally — Prenatally: pills by mouth, one per day, from the first prenatal visit until delivery, 400 mcg folic acid.
  Postnatally: liquid by mouth, once per day, from 6 weeks old until 9 months old, 1 mg/kg/day Fe, 1500 IU vitamin A, 500 IU vitamin D.
  Arms: c
Dietary Supplement: folic acid prenatally, vitamins A & D postnatally — Prenatally: pills by mouth, one per day, from the first prenatal visit until delivery, 400 mcg folic acid.
  Postnatally: liquid by mouth, once per day, from 6 weeks old until 9 months old, 1500 IU vitamin A, 500 IU vitamin D.
  Arms: d

SUMMARY:
The Healthy Infant Development Project will determine if providing micronutrient supplements to mothers during pregnancy and infants in the first 9 months fosters healthy behavior and development in babies.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the most common single nutrient disorder in the world, and pregnant women and infants are at highest risk. With long-lasting differences in prior studies, effects on the developing brain and infant behavior and development are among the most worrisome concerns. The proposed study will determine developmental/ behavioral effects of preventing ID depending on timing (Aim 1) and duration (Aim 2) of iron supplementation (i.e., pre- and/or early postnatally). The study will relate outcomes to severity of ID (Aim 3) and consider reversibility of effects with iron therapy, depending on timing (Aim 4). We expect different neurobehavioral effects when ID occurs or is prevented/treated during different phases of brain development (proliferation and growth phase primarily prenatally and regional diversification and interconnection largely in infancy). The project entails 2 randomized controlled trials (RCTs) to support causal inferences about preventing ID pre- and/or early postnatally. The project builds on a large US CDC-supported study (Pregnancy Nutrition Study) involving pregnant women in rural China (ClinicalTrials.gov identifier: NCT00133744). Study groups of infants in the proposed RCTs combined are a) pre- and early postnatal iron, b) prenatal iron, c) early postnatal iron, and d) neither (n = 500/group, total 2000, at study end). Iron status and sensitive sensory, motor, cognitive, language, and social-emotional outcomes will be assessed at birth, 9 and 18 mo. Results of Aims 1 & 2 will determine the best window to prevent ID effects and whether breast-fed infants benefit from iron before 6 mo. Aim 3 (severity) will determine the level of ID at which different developmental domains are adversely affected. If ill effects of ID without anemia are documented, there could be major policy implications; screening is currently only for anemia. Detecting more or less vulnerable domains may also point to other interventions in addition to iron therapy. To identify reversibile effects, depending on age of treatment (Aim 4), outcomes at 18 mo will be compared for infants 1) never iron-deficient, 2) poor iron status at birth and assigned to postnatal iron, 3) maternal IDA (anemia) treated in the 1st or 2nd trimester, 4) infant IDA treated at 9 mo, and 5) IDA treated at 18 mo. The results will be highly relevant to global practice and policy regarding ID, which differentially affects poor and/or minority women and infants everywhere.

The project is expected to continue with a 5-year follow-up (Nov 2014- Oct 2019).

ELIGIBILITY:
Inclusion Criteria:

- Full-term healthy neonates born to study mothers from CDC's Prenatal Nutrition Study with randomly selected lot numbers.

Exclusion Criteria:

* birth weight < 2500 g
* gestational age ≤ 37 wk
* major perinatal complications
* major congenital anomaly
* multiple birth.

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2371 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Infant behavior and development | 9 and 18 months

SECONDARY OUTCOMES:
Infant anemia | 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lozoff, MD, Principal Investigator — University of Michigan; Li Ming, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Clark KM, Li M, Zhu B, Liang F, Shao J, Zhang Y, Ji C, Zhao Z, Kaciroti N, Lozoff B. Breastfeeding, Mixed, or Formula Feeding at 9 Months of Age and the Prevalence of Iron Deficiency and Iron Deficiency Anemia in Two Cohorts of Infants in China. J Pediatr. 2017 Feb;181:56-61. doi: 10.1016/j.jpeds.2016.10.041. Epub 2016 Nov 8. PMID 27836288
- [Derived] Lozoff B, Jiang Y, Li X, Zhou M, Richards B, Xu G, Clark KM, Liang F, Kaciroti N, Zhao G, Santos DC, Zhang Z, Tardif T, Li M. Low-Dose Iron Supplementation in Infancy Modestly Increases Infant Iron Status at 9 Mo without Decreasing Growth or Increasing Illness in a Randomized Clinical Trial in Rural China. J Nutr. 2016 Mar;146(3):612-21. doi: 10.3945/jn.115.223917. Epub 2016 Jan 20. PMID 26791556